CLINICAL TRIAL: NCT00099580
Title: PROCLAIM: A Phase 2, Randomized, Double-Blind, Parallel-Group, Placebo-Controlled, Multicenter Study to Examine the Effects of AC2592 Administered by Continuous Subcutaneous Infusion in Subjects With Advanced Chronic Congestive Heart Failure
Brief Title: PROCLAIM: Effect of AC2592 Administered by Continuous Subcutaneous Infusion in Subjects With Advanced Chronic Congestive Heart Failure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2592-101 (PROCLAIM)
Record Dates: First submitted 2004-12-17; First posted 2004-12-20 (Estimated); Last update posted 2015-01-19 (Estimated); Status verified 2014-12

CONDITIONS: Congestive Heart Failure
Keywords: Congestive Heart Failure; AC2592; GLP-1; Amylin; metabolic abnormality
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: AC2592
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: AC2592 — continuous subcutaneous infusion (via pump), dose based on subject body weight
  Arms: 1
Drug: placebo — continuous subcutaneous infusion (via pump), dose based on subject body weight
  Arms: 2

SUMMARY:
This Phase 2, randomized, placebo-controlled, multicenter outpatient study is designed to test the safety and tolerability of AC2592 as well as examine the effect of AC2592 on oxygen consumption during maximal tolerated exercise in adult subjects with chronic congestive heart failure.

ELIGIBILITY:
Main Inclusion Criteria:

* Has heart failure classified as New York Heart Association (NYHA) Class III or Class IV at screening despite treatment with standard therapy.
* Is able to perform a treadmill test.
* Has an HbA1c of <= 11%.
* Is physically and mentally capable of operating the continuous subcutaneous infusion (CSCI) pump (i.e., adequate vision, manual dexterity, and mental capacity), or has a dedicated caretaker or adult family member who meets this requirement.

Main Exclusion Criteria:

* Has received metformin or nesiritide within 2 weeks prior to screening visit.
* Is currently participating in any other clinical study, or has received an investigational drug within 1 month of the screening period.
* Has participated previously in a study using GLP-1, exenatide, or exenatide LAR.
* Is using a left ventricular assist device or other mechanical circulatory support.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2005-03; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
To examine the safety and tolerability of AC2592 administered by continuous subcutaneous infusion in subjects with chronic congestive heart failure. | 6 weeks
To assess the effect of AC2592 administered by continuous subcutaneous infusion on oxygen consumption during maximal tolerated exercise in adult subjects with chronic congestive heart failure. | 6 weeks

SECONDARY OUTCOMES:
To assess the effect of AC2592 administered by continuous subcutaneous infusion on pharmacokinetics, pharmacodynamics, and clinical outcomes in adult subjects with chronic congestive heart failure. | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Porter, MD, Study Director — Amylin Pharmaceuticals, LLC.
Locations (29):
- United States (29):
  - Research Site, Beverly Hills, California
  - Research Site, Mission Viejo, California
  - Research Site, New Haven, Connecticut
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Jacksonville, Florida
  - Research Site, Tampa, Florida
  - Research Site, Peoria, Illinois
  - Research Site, Springfield, Illinois
  - Research Site, Winfield, Illinois
  - Research Site, Wichita, Kansas
  - Research Site, Baton Rouge, Louisiana
  - Research Site, Shreveport, Louisiana
  - Research Site, Auburn, Maine
  - Research Site, Boston, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, Lincoln, Nebraska
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Durham, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Medford, Oregon
  - Research Site, Portland, Oregon
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Charleston, South Carolina
  - Research Site, Knoxville, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas